CLINICAL TRIAL: NCT06886022
Title: The Establishment of a Diagnosis, Treatment, and Prevention System for Colorectal Cancer Under the Background of Abnormal Lipid Metabolism in Digitalization
Brief Title: Diagnosis, Treatment, and Prevention of Colorectal Cancer Amid Abnormal Lipid Metabolism
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Union Medical Center (Other)
Responsible Party: Principal Investigator, Jing Xu, Chief Physician, Tianjin Union Medical Center
Other Study IDs: 2023C03
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Lipid Metabolism
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum; Adipose Tissue; Tumor tissue; Skeletal Muscle tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation: Colorectal cancer patients after surgery
  Interventions: Procedure: Colorectal cancer procedures

INTERVENTIONS:
Procedure: Colorectal cancer procedures — Procedures

SUMMARY:
This research project investigates the interplay between lipid metabolism, inflammation, and colorectal cancer (CRC). We are building a comprehensive database of CRC patients, incorporating clinical data, body composition measurements, imaging findings, and biomarkers related to lipid metabolism and inflammation. Our goal is to identify how these factors contribute to CRC development, progression, and perioperative outcomes. Ultimately, we aim to develop a digital, personalized "three-tier prevention" strategy encompassing early risk prediction, targeted interventions, and comprehensive rehabilitation for improved CRC patient care.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common gastrointestinal malignancies worldwide, accounting for approximately 8% of all cancer cases [1]. Numerous epidemiological studies have identified obesity as a risk factor for CRC [2]. Abnormal fat distribution and lipid metabolism dysregulation contribute to a chronic, low-grade inflammatory state and increased oxidative stress, potentially triggering mutations, carcinogenesis, and tumor cell proliferation [3]. Research suggests that adipose tissue and its associated inflammatory factors may play a key role in the obesity-cancer link.

Regarding fat distribution, visceral adipose tissue exhibits higher metabolic activity compared to subcutaneous fat [4]. Excess visceral fat promotes insulin resistance and inflammatory pathways [5], potentially increasing CRC risk. Abnormal visceral fat distribution is also associated with postoperative complications, survival time, and the efficacy of adjuvant therapy in CRC patients [6]. Furthermore, non-alcoholic fatty liver disease (NAFLD), potentially representing a specific type or hepatic manifestation of abnormal fat distribution, is considered a risk factor for CRC.

Our research group previously conducted a retrospective study involving 93 patients undergoing gastrointestinal surgery (including CRC). We found that, compared to the group without perioperative weight loss, patients experiencing perioperative weight loss exhibited decreased serum albumin, elevated blood glucose, and elevated serum cholesterol. Multivariate regression analysis indicated that serum cholesterol was a risk factor for perioperative weight loss, showing a positive correlation.

Currently, we are conducting a small-scale study specifically focusing on CRC patients. By collecting perioperative data, including body composition, fat distribution, BMI, abdominal CT scans, inflammatory markers, and obesity-related indices, we aim to elucidate the roles of lipid metabolism, fat distribution, and related inflammatory factors in the development and progression of CRC, as well as their impact on perioperative adverse clinical outcomes. We have obtained promising preliminary results, establishing a foundation for digitizing our overall research findings.

This project aims to establish a research system correlating lipid metabolism, inflammation, and CRC. A CRC patient lipid metabolism database will serve as a platform to expand our previous study's sample size. By integrating and analyzing data from this platform, we will develop a digital, visualized "three-tier prevention" network for CRC, integrating a "digital vaccine" (predictive screening model), "digital drug" (intervention model targeting associated pathogenic mechanisms), and "digital rehabilitation" (preventive system combining early warning and treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years, confirmed CRC diagnosis, consent to participate in the study.

Exclusion Criteria:

* Age <20 or >80 years; inability to perform activities of daily living; presence of infectious diseases; lack of communication and cognitive abilities; refusal to participate in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 20-80 years, confirmed CRC diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal CT L3 level adipose tissue surface | Preoperatively
  Abdominal CT L3 level adipose tissue surface
Abdominal CT L3 level skeletal muscle surface | Preoperatively

SECONDARY OUTCOMES:
Tumor TNM stage | immediately after the procedure
Overall Survival | 3 years
Disease Free Survival | 3 years
Hand grip strength | Preoperatively; Postoperatively Day 1,3,5,7
Waist Circumference | Preoperatively
Calf Circumference | Preoperatively; Postoperatively Day 1 3 5 7
Progression Free Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xu, PhD, Principal Investigator — Tianjin Union Medical Center

IPD SHARING:
Plan to Share IPD: No